CLINICAL TRIAL: NCT00266773
Title: Therapeutic Interactive Voice Response (IVR) for Relapse Prevention in Chronic Pain
Brief Title: A Telephone Feedback System for Prevention of Chronic Pain Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Magdalena Naylor, MD, PhD, Magdalena R. Naylor, MD, PhD, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR052131 (NIH); R01AR052131 (NIH); 5R01AR052131 (NIH)
Record Dates: First submitted 2005-12-16; First posted 2005-12-19 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Pain and Relapse Prevention
Keywords: Chronic Pain; Cognitive Therapy; Cognitive Behavioral Therapy; Recurrence; Relapse Prevention; Educational Technology; CBT; CST; IVR; TIVR
MeSH Terms: conditions — Chronic Pain; Recurrence | interventions — Drug Delivery Systems

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (No Intervention): Control - standard care only
- 2 (Experimental): Attention Control - standard care plus 6 months TIVR receiving minimal monthly feedback
  Interventions: Behavioral: Chronic pain therapeutic interactive voice response (TIVR) system
- 3 (Experimental): Standard care plus 6 months TIVR receiving detailed monthly feedback
  Interventions: Behavioral: Chronic pain therapeutic interactive voice response (TIVR) system

INTERVENTIONS:
Behavioral: Chronic pain therapeutic interactive voice response (TIVR) system — Therapeutic Interactive Voice Response as a daily self monitoring and relapse prevention tool with didactic reviews and practices of recorded skills and monthly feedback based on daily calls
  Arms: 2; 3

SUMMARY:
The purpose of this study is to determine whether a telephone-based self-monitoring and skills review program with personalized therapist feedback following group CST for chronic pain can reduce and prevent relapse of the pain, physical disability, and psychological distress experienced by patients with chronic pain of the muscles and bone.

DETAILED DESCRIPTION:
IVR (Interactive Voice Response) is a computer-based, automated telephone system that enables callers to respond to a recorded voice via the telephone keypad. Using this technology, therapeutic IVR (TIVR) was developed as a tool for providing maintenance treatment following group cognitive-behavioral coping skills training (CST), a widely-used behavioral treatment for chronic pain. TIVR has four components:

* an automated daily questionnaire for self-monitoring
* a review of coping skills
* guided behavioral rehearsals of CST coping skills
* personalized monthly feedback messages recorded onto TIVR by the therapist

All four components can be accessed remotely by patients via any touch-tone phone. In a small pilot study, people with severe, chronic musculoskeletal pain received 11 weeks of either CST alone or CST with TIVR access and therapist feedback. Those who used TIVR had better pain outcomes than those who did not. This study will compare the effectiveness of TIVR with or without therapist feedback to a control group not using TIVR at all.

To be eligible for this study, participants must have just completed an 11-week course of CST through the University of Vermont College of Medicine's MindBody Medicine Clinic. At study entry, participants will be randomly assigned to one of three groups. Group 1 is a control group that will not receive any intervention through this study. Group 2 participants will receive full access to TIVR and will get a minimal monthly message from their therapist, who will not use the participant's daily questionnaire data. Group 3 participants will receive full access to TIVR and will get personalized monthly messages from their therapist based on the participant's daily questionnaire data. Messages for participants will include any trends the therapist has noted in a participant's stress, sleep, mood, pain levels, coping, and activity, as reported through TIVR. All study participants may continue to receive treatment from their regular physician or take part in other pain management techniques during this study, but such treatment will not be provided through this study.

Upon completing the 11 weeks of CST, all participants will be asked to complete a packet of questionnaires about their chronic pain. At the start of this study, participants in Groups 2 and 3 will have a 30-minute training session on how to use and access TIVR. At Months 4, 8, and 12, participants from all three groups will have follow-up interviews and will complete additional questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Completed 11 weeks of CST through the University of Vermont College of Medicine - Health Behavior Research Center prior to study entry
* At least 6 months of musculoskeletal pain caused by back, neck, or shoulder pain; osteoarthritis; or fibromyalgia
* Meet study threshold for pain severity with a Typical Pain score of 4 or more on a 10-point scale adapted from the McGill Pain Questionnaire (80)
* Receiving ongoing standard pain management from a physician (typically involving oral analgesic medication and physical therapy, with or without anesthetic or steroid injections)

Exclusion Criteria:

* Unable to perform usual self care
* Cancer that causes or influences patient's chronic pain
* Cancer requiring radiation or chemotherapy or metastatic cancer of any type
* Reflex sympathetic dystrophy (RSD)
* Neuropathic pain
* Awaiting a pain-related surgical procedure
* Involved in pain-related litigation or awaiting disability determination
* Behavioral problems or psychotic disorders that may interfere with the study
* Inability to use telephone-based TIVR due to cognitive or hearing impairment
* At risk for suicide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2005-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Total pain experience and physical and social disability (as measured by the TOPS) | 12 months
Pain level (as measured by the McGill Pain Questionnaire) | 12 months
Catastrophizing and perceptions of control (as measured by the Coping Strategies Questionnaire) | 12 months

SECONDARY OUTCOMES:
Utilization of telephone system components during the study | daily for 6 months
Daily ratings of mood, pain, and coping use (measured by the TIVR Daily Questionnaire) | daily for 6 months
General measure of depressive symptoms (measured by the Beck Depression Inventory) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena R. Naylor, MD, PhD, Principal Investigator — University of Vermont College of Medicine - MindBody Medicine Clinic
Locations (1):
- University of Vermont College of Medicine - MindBody Medicine Clinic, Burlington, Vermont, United States

REFERENCES:
- [Background] Keefe FJ, Rumble ME, Scipio CD, Giordano LA, Perri LM. Psychological aspects of persistent pain: current state of the science. J Pain. 2004 May;5(4):195-211. doi: 10.1016/j.jpain.2004.02.576. PMID 15162342
- [Background] Naylor MR, Helzer JE, Naud S, Keefe FJ. Automated telephone as an adjunct for the treatment of chronic pain: a pilot study. J Pain. 2002 Dec;3(6):429-38. doi: 10.1054/jpai.2002.129563. PMID 14622728
- See also: Click here for the University of Vermont College of Medicine - MindBody Medicine Clinic Web site — http://www.med.uvm.edu/mbmc